CLINICAL TRIAL: NCT05102994
Title: The Diagnostic Value of Mutation Detection for VRL
Brief Title: Mutation Detection for VRL
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Dan Liang, PhD, Sun Yat-sen University
Other Study IDs: 2021-VRL-diagnosis
Record Dates: First submitted 2021-10-17; First posted 2021-11-02 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Vitreoretinal Lymphoma; Uveitis
Keywords: Vitreoretinal lymphoma; Uveitis; intraocular fluid; mutation
MeSH Terms: conditions — Intraocular Lymphoma; Uveitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Combined ocular manifestations with the results of pathology, IL-10/IL-6 ratio, IGH gene rearrangements and patients' response to treatments, patients abtained clear diagnosis
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- VRL patients group: Presenting clinical features suggestive for VRL with positive finding in laboratory exam
  Interventions: Diagnostic Test: mutation test
- uveitis group: Even if characterized as clinical features of presumed VRL, no positive laboratory investigations for lymphoma and well response to IMT
  Interventions: Diagnostic Test: mutation test

INTERVENTIONS:
Diagnostic Test: mutation test — detect the tumor-related mutation in introcular fluid

SUMMARY:
Vitreoretinal lymphoma (VRL) is a rare but aggressive masquerade syndrome, which would be easily confused with uveitis. The diagnostic gold standard remains the pathologic examination of ocular specimen with invasiveness and low sensitivity. To improve the safety and accuracy of VRL diagnosis, alternative techniques using intraocular fluid (IOF) samples are emerging. In this study, we aimed to test the diagnostic value of mutation analysis for VRL

DETAILED DESCRIPTION:
chest CT, urinalysis, kidney, and liver function were routinely checked.

IL-10/IL-6 ratio, genetic mutation analysis and samples were IGH gene rearrangements were reviewed and analyzed retrospectively.

The diagnoses were identified after careful evaluation of treatment effects in follow-up. The diagnostic value including sensitivity, specificity, positive and negative predictive values, and test efficiency of genetic mutation analysis in diagnosing VRL were analyzed.

Furthermore, a validation group of patients including VRL and uveitis was selected to validate the diagnostic value of mutation analysis in the diagnosis of VRL. All the patients signed an informed consent and institutional review board approval was obtained. The study was performed in accordance with the tenets of the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* suspected VRL patients who had intraocular fluid for mutation test. And got a clear diagnose of VRL or uveitis afther having dianostic tests and follow-up treatment

Exclusion Criteria:

* suspected VRL patients who lost in follow-up without a definitive diagnose, or whoever reluctance to participate our study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: suspected VRL or uveitis patients attending to our clinic
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-11-10 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
the result of mutation test | at baseline, before treatment
  any mutation detect in intraocular fluild recorded as ctDNA+

CONTACTS AND LOCATIONS:
Overall Officials: Dan D Liang, PhD, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No